CLINICAL TRIAL: NCT01019759
Title: The Value of add-on Arrhythmia Surgery in Patients With Paroxysmal or Persistent Atrial Fibrillation Undergoing Valvular or Coronary Bypass Surgery. A Randomised Comparison on Quality of Life, Cost-effectiveness, Morbidity and Rhythm Outcome.
Brief Title: The Value of add-on Arrhythmia Surgery in Patients With Atrial Fibrillation Undergoing Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Prof Dr. JG Maessen, dept Cardiothoracic Surgery, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MEC 02-119.3; PF 178
Record Dates: First submitted 2009-07-06; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; cardiac surgery; ablation; pulmonary veins
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No add-on AF-surgery (No Intervention): patient undergoing only scheduled valve and/or coronary bypass surgery
- PV isolation (Experimental): patient undergoing add-on epicardial microwave energy pulmonary vein isolation
  Interventions: Procedure: pulmonary vein isolation

INTERVENTIONS:
Procedure: pulmonary vein isolation — The off-pump beating heart ablation procedure is performed. Using a Microwave (MW) energy ablation tool (Microwave generator by Guidant), epicardial ablation line isolating the pulmonary veins are applied during open heart surgery
  Other Names: Microwave generator by Guidant; Flex 4 or Flex 10 ablation probes by Guidant
  Arms: PV isolation

SUMMARY:
The hypothesis being studied is that add-on arrhythmia surgery in patients with atrial fibrillation (AF) undergoing valvular or coronary surgery improves quality of life, is cost-effective, reduces perioperative and long-term morbidity associated with AF.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is connected with an increased morbidity and mortality. In addition, quality of life is diminished due to palpitations, dyspnea, dizziness and syncope. AF is frequently associated with valvular and coronary disease. In the AF patients undergoing valvular or coronary surgery the arrhythmia almost always relapses. For symptom control anti-arrhythmic drugs and cardioversion are used but breakthrough arrhythmias and side effects of the drugs happen frequently. For more effective symptom control "add-on" arrhythmia surgery is being advocated. However, at present we do not know whether add-on arrhythmia surgery indeed affects morbidity and quality of life. In this respect the benefit of chronic sinus rhythm has to outweigh the risks of a prolonged operation. In addition, cardiovascular complaints unrelated to AF may persist even after successful operation, thus offsetting the benefit of chronic sinus rhythm. Add-on surgery is more costly than standard surgery but this may compare favourably with shorter hospital admission due to less frequent post-operative AF.

Valvular heart disease is frequently associated with ventricular remodelling: a decreased ventricular function and atrial dilatation. AF itself may worsen heart failure due to a tachycardiomyopathy. Elimination of AF might therefore enhance recovery from structural and functional remodelling and promote recovery of quality of life after the operation.

The PIAF, RACE and AFFIRM have shown that chronic sinus rhythm is not necessarily associated with a reduced morbidity or enhanced quality of life. PIAF however showed that exercise tolerance was better when rhythm control was achieved. Further analyses of RACE and AFFIRM are pending. One drawback of the above studies is the fact that chronic sinus rhythm is difficult to obtain. In PIAF, RACE and AFFIRM only 30 to 50% was in sinus rhythm at the end of follow-up. By contrast, arrhythmia surgery is a highly effective treatment in this respect.

Forty patients underwent a (phase 1-study) coronary bypass- or valve surgery with add-on arrhythmia surgery in the same way as in this protocol proposed. This means epicardial on beating heart and without use of the heart-lung machine. In the last follow-up 80 % of the patients not longer were in atrial fibrillation. With similar treatment procedures, but more invasive, so on the arrested heart and endo cardially, success percentages reported varying from 60 % till 80%.

This large variance in success rate is probably related to the primary course of the disease and the degree of the morphological abnormality. In spite of these meaningful results ''add-on'' arrhythmia surgery is no general accepted treatment. The intended patient population remains generally untreated. Historical data of patients from the university hospital of Maastricht show that no add on treatment has a success rate of 25% of patients in sinus rhythm.

Considering the above a randomised comparison of add-on arrhythmia surgery and standard surgery is warranted.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergo valvular surgery, coronary surgery, or a combination of both.
2. All patients have documented chronic atrial fibrillation of paroxysmal atrial fibrillation.
3. Patients have given written informed consent.

Exclusion Criteria:

1. Patients who do not speak Dutch or can not read Dutch.
2. Patients with a Sick Sinus Syndrome.
3. Patients with contraindications for oral anticoagulant agents.
4. Patients unable to express their specific wishes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2002-09; Primary Completion 2006-11 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients free from atrial fibrillation, as apparent from 24 hour Holter registration, in addition to standard ECG. For the purpose of this primary endpoint, AF was defined as lasting longer than 10 seconds. | between 3 months and 12 months post-operative

SECONDARY OUTCOMES:
Quality of life (QoL) | at 3, 6 and12 months post-operative
Cost-effectiveness | intraoperative untill 12 months post-operative
In-hospital morbidity (incl. pulmonary complications, resternotomy for surgical bleeding, cerebrovascular accidents, acute myocardial infarction, renal failure, development of atrioventricular conduction abnormalities) | post-operative, in-hospital period
Rhythm related events and interventions (incl. electrical or chemical cardioversion, percutaneous catheter ablation, implantation of a defibrillator, pacemaker implantation) | discharge untill 12 months post-operative
Out-of-hospital morbidity (incl. acute myocardial infarction, percutaneous catheter ablation, implantation of a defibrillator, pacemaker implantation and cerebrovascular accidents, syncope) | discharge untill 12 months post-operative
Mortality | intraoperative untill 12 months post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Jos G Maessen,, MD, PhD, Principal Investigator — dept. Cardiothoracic Surgery, University hospital of Maastricht
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands